CLINICAL TRIAL: NCT06546241
Title: Celebrándome: A Body Confidence Program for Hispanic/Latinx Youth
Brief Title: Celebrandome: Preliminary Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Dove Self Esteem Project, Unilever Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00017437
Record Dates: First submitted 2023-03-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Body Image; Self Esteem

STUDY DESIGN:
Intervention Model Description: Participants are randomized to the intervention or wait-list control group. The intervention group will complete a baseline survey, receive the 60 minute workshop, and completes a post-intervention survey. The control group receives a survey, waits, completes a baseline survey, then receives the 60 minute workshop, and completes a post-intervention survey.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The project coordinator and PI oversee the randomization and participant tracking. However, participants do not know their assigned condition, and facilitators that run the workshops are blind to participant condition, and undergraduate research assistants that oversee the distribution of surveys are blind to participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Hispanic/Latinx youth between the ages of 11 to 16 will participate in a 60 minute workshop aimed and increasing body image satisfaction and self esteem. Participants randomized to the intervention group are scheduled immediately to receive the intervention. The intervention is delivered in a group format with groups consisting of no more than 20 youth.
  Interventions: Behavioral: Celebrandome
- Wait-List Control Group (No Intervention): The control group is a waitlist control group. Participants in the control group complete a survey, wait for 2 to 3 weeks, then are eligible to sign up for the workshop. During the wait-list period they complete 2 surveys.

INTERVENTIONS:
Behavioral: Celebrandome — This intervention is based on existing cognitive dissonance body confidence programs for youth such as Amazing Me, Free Being Me, and Body Project. Consistent with these programs, workshops are entirely experiential getting you to discuss appearance ideals and why they are problematic, pressures they experience to conform to appearance ideals, ways to combat pressures, they compare pictures that are normal versus digitally altered and discuss ways this is problematic, they discuss body talk statements they hear all the time and how this promotes appearance ideals, they practice ways to combat body talk statements. They develop positive affirmation statements. In addition and unique to this curriculum, all activities highlight cultural ideals and how youth can receive different messages related to different appearance ideals and they unique stress and pressures this creates.
  Other Names: Body Confidence Single Session
  Arms: Intervention Group

SUMMARY:
The Dove Self Esteem Project, has provided our research team with funding to develop a 60- minute workshop for Hispanic/Latinx Youth between the ages of 11 to 16 years old that builds body confidence. This workshop was developed based on prior curriculum the investigator has developed for The Dove Self Esteem Project and designed with two teachers and several adolescent children.

The aims of the current study are to: 1) examine the efficacy of the workshop, and 2.) evaluate the extent to which children like the curriculum and find it useful. Children will be randomized to control group or intervention group; however, the control group will eventually go through the workshop after 2 surveys. It is hypothesized that children in the intervention group will report higher body satisfaction scores, greater self- esteem, more awareness of body talk and less engagement in appearance comparisons relative to the control group. It is hypothesized that children will report liking the workshop, finding it useful and engaging.

ELIGIBILITY:
Inclusion Criteria:

* Youth who are 11 to 16 years of age
* Youth who identify as Hispanic/Latino/Latinx
* Youth who are fluent in English

Exclusion Criteria:

* None.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Baseline - Body Image Self Esteem (Body Esteem Scale; Mendelson & White, 1982) | This measure is administered immediately before the intervention.
  This measure assesses the extent youth like their appearance and the extent they dislike their appearance. Higher scores indicate more self esteem. Instructions are "Right now, please tell us how much this represents you." Items are on a Likert scale from 0 (never) to 4 (Always).
Post - Body Image Self Esteem (Body Esteem Scale; Mendelson & White, 1982) | This measure is administered immediately after the intervention.
  This measure assesses the extent youth like their appearance and the extent they dislike their appearance. Higher scores indicate more self esteem. Instructions are "Right now, please tell us how much this represents you." Items are on a Likert scale from 0 (never) to 4 (Always).
Baseline - General Self Esteem (Rosenberg Self-Esteem Scale - Child Version; -Rosenberg, 1965) | This measure is administered immediately before the intervention.
  This measure assesses the extent to which a person like themselves or feels competent. Higher scores indicate more higher self esteem. Instructions are "Right now, please tell us how much this represents you." Items are on a Likert scale from 0 (I strongly agree ) to 3 (I strongly disagree).
Post - General Self Esteem (Rosenberg Self-Esteem Scale - Child Version; Rosenberg, 1965) | This measure is administered immediately after the intervention.
  This measure assesses the extent to which a person like themselves or feels competent. Higher scores indicate more higher self esteem. Instructions are "Right now, please tell us how much this represents you." Items are on a Likert scale from 0 (I strongly agree ) to 3 (I strongly disagree).

SECONDARY OUTCOMES:
Baseline - Appearance Conversations Scale (Jones, Vigfusdottir, & Lee, 2004). | This measure is administered immediately before the intervention.
  This measure assesses the extent a youth talks about appearance with friends. Instructions are "how often do you talk about the following things with your friends?" Items are on a Likert scale form 0 (never) to 4 (very often), with higher scores indicating higher frequency of engaging in appearance conversations.
Post - Appearance Conversations Scale (Jones, Vigfusdottir, & Lee, 2004). | This measure is administered immediately after the intervention.
  This measure assesses the extent a youth talks about appearance with friends. Instructions are "how often do you talk about the following things with your friends?" Items are on a Likert scale form 0 (never) to 4 (very often), with higher scores indicating higher frequency of engaging in appearance conversations.
Baseline - Pressures to Conform to Appearance Ideals (Sociocultural Pressures Scale; Diedrichs, Atkinson, Steer, 2015) | This measure is administered immediately before the intervention.
  Assesses how often children feel pressure from friends, family or the media to change different aspects of their appearance. Instructions are "please circle how often you do this..." Items are on a Likert scale from 0 (none) to 4 (a lot), with higher scores indicating more feeling more pressure.
Post - Pressures to Conform to Appearance Ideals (Sociocultural Pressures Scale; Diedrichs, Atkinson, Steer, 2015) | This measure is administered immediately after the intervention.
  Assesses how often children feel pressure from friends, family or the media to change different aspects of their appearance. Instructions are "please circle how often you do this..." Items are on a Likert scale from 0 (none) to 4 (a lot), with higher scores indicating more feeling more pressure.
Baseline - Appearance Comparisons (Social Comparison to Models and Peers Scale; Jones, 2001) | This measure is administered immediately before the intervention.
  Assesses how often children compare themselves to kids their age or celebrities/people in the media. Instructions are "lease circle how often you do this..." Items are on a Likert scale from 0 (never) to 4 (a lot), with higher scores indicating more engagement in appearance comparisons.
Post - Appearance Comparisons (Social Comparison to Models and Peers Scale; Jones, 2001) | This measure is administered immediately after the intervention.
  Assesses how often children compare themselves to kids their age or celebrities/people in the media. Instructions are "lease circle how often you do this..." Items are on a Likert scale from 0 (never) to 4 (a lot), with higher scores indicating more engagement in appearance comparisons.

OTHER OUTCOMES:
Palatability Characteristics of the Program | Assessed in the intervention condition only, immediately after the workshop.
  Assesses the extent youth enjoy, understand, feel comfortable with the workshop. Instructions are "Right now, tell us your thoughts on the workshop you just participated in."

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Pending IRB approval, researchers can contact the PI to obtain the de-identified data.